CLINICAL TRIAL: NCT06452407
Title: Evaluating the Feasibility of elleFA App Implementation
Acronym: elleFA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Andrew Zakhari, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2025-10774
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-09

CONDITIONS: Endometriosis
Keywords: mobile health application; app; symptom tracking; treatment tracking; self-tracking; pain; quality of life; patient-provider communication
MeSH Terms: conditions — Endometriosis; Alzheimer Disease; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implementation of elleFA smartphone application (Experimental): Implementation of the elleFA smartphone application to track symptoms, lifestyle, treatments and any patient-defined endpoints.
  Interventions: Other: Implementation of elleFA smartphone application

INTERVENTIONS:
Other: Implementation of elleFA smartphone application — Participants will download the elleFA application on their smartphone. Through this application, the user will be prompted to complete a short modified Biberoglu and Behrman (B&B) questionnaire and a longer EHP-30 questionnaire monthly, for a period of 6 months. Optionally, patients may complete an additional weekly summary of their mental health symptoms, pain localization, and other symptoms. Also optionally, they may record any daily symptoms, separated into categories from lifestyle to physical pain, objectified through a 5-point Likert scale.

SUMMARY:
Endometriosis is a chronic incurable disease where endometrial-like tissue grows outside of the uterus, and causes symptoms such as debilitating menstrual pain, pain during intercourse, infertility, constipation, and bloating, which hurts their quality of life. Endometriosis is estimated to affect approximately 10% of women. Despite this, there's currently not enough research on this disease; in Canada it takes on average 5.4 years to get a diagnosis (from when symptoms start), and once diagnosed, women often have to go through a trial-and-error process to find a treatment that can manage their symptoms. Misunderstanding symptoms and struggling with patient-provider communication both contribute to these delays in diagnosis and finding the best treatment.

Mobile health applications have been a promising new tool to self-track symptoms and treatments. There are several apps currently available on the market for logging chronic pain, menstrual cycles, and fertility. However, no apps exist specifically for endometriosis that look at the whole spectrum of symptoms, including pain, quality of life, and especially ease of patient-provider communication. The elleFA app is a new, personal endometriosis and health tracking app designed to improve patient-physician dialogue through more direct, efficient, and impactful communication, as patients navigate their condition.

This single-arm interventional study aims to test the feasibility of implementing the new elleFA app in a clinical setting for 6 months in pre-menopausal women 18 years and older with endometriosis, and the app's impact on patient experience. Participants will download the elleFA app on their smartphone and will be asked to complete two questionnaires through the app every month for 6 months. Participants can choose to also optionally track their daily symptoms, lifestyle, and treatments, through weekly symptom log summaries through the app.

The main study finding will be be patient adherence to using the app over a 6 month study period. Other findings will include user-reported satisfaction with the elleFA app, and the impact of elleFA app use on patient experience communicating with their healthcare team.

DETAILED DESCRIPTION:
Endometriosis is a chronic incurable disease where endometrial-like tissue grows outside of the uterus and is estimated to affect 10% of women of reproductive age. Many women with endometriosis experience symptoms including but not limited to debilitating menstrual pain, pain during intercourse, infertility, constipation, and bloating. Their quality of life is severely hindered, with an average of 0.809 quality-adjusted life years per woman suffering from the condition. Endometriosis is currently deeply under-researched; diagnosis is delayed on average 5.4 years from the onset of symptoms in Canada, and once diagnosed, women often have to undergo a trial-and-error approach to find treatment strategies to manage their symptoms. Misunderstanding symptoms for common menstrual pains as well as struggles in patient-provider communication in the form of physician dismissal or patient recall bias and memory gaps contribute to these delays in diagnosis and appropriate treatments.

Mobile health applications have been a promising new tool to self-track symptoms and treatments. Women report being motivated to use this mode of tracking to better manage their symptoms and improve communication with their healthcare providers. There are several apps currently available on the market for logging chronic pain, menstrual cycles, and fertility. However, endometriosis patients report feeling limited by these apps, as no apps exist specifically for endometriosis that look at the whole spectrum of symptoms, including pain, quality of life, and especially ease of patient-provider communication. Therefore, in this pilot study, we propose determining the feasibility of introducing the novel elleFA app in the clinical setting, a personal endometriosis and health tracking app designed to improve patient-physician dialogue through more direct, efficient, and impactful communication, as patients navigate their condition.

This 6-month prospective open-label single-arm interventional clinical study aims to test the feasibility of implementing the elleFA app for 6 months in women with endometriosis, and its impact on patient experience. Twenty pre-menopausal women 18 years or older with suspected or confirmed endometriosis will be recruited. Upon recruitment, each participant will fill out a brief demographic questionnaire, then download the elleFA app on their smartphone and will be asked to complete two validated questionnaires monthly, for 6 months. Daily symptom, lifestyle, and treatment tracking, as well as weekly symptom log summaries, are available for optional completion by the participant.

The primary outcome will be patient adherence to using the app as defined by the completion rate of monthly modified Biberoglu and Behrman (B&B) scale and Endometriosis Health Profile (EHP-30) surveys over a 6 month study period. One secondary outcome will be reported user satisfaction with the elleFA app itself, measured by score of patient-reported questionnaire designed to capture the user experience and perceived app functionality using a 5-point Likert scale. Another secondary outcome will be the impact of elleFA app use on patient experience communicating with the healthcare team, measured by factors such as confidence in recall or comfort with the physician-patient relationship using a 5-point Likert scale.

ELIGIBILITY:
Inclusion Criteria:

* Pre-menopausal women 18 years of age or older with known or suspected endometriosis
* Undergoing medical management of endometriosis at the MUHC
* Able to provide informed consent in French or in English

Exclusion Criteria:

* Menopausal status
* Pregnant or seeking pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
patient adherence to using the app | 6-months following trial commencement
  Completion rate of monthly modified Biberoglu and Behrman (B&B) scale and Endometriosis Health Profile (EHP-30) surveys over a 6 month study period, retrieved electronically.

SECONDARY OUTCOMES:
Patient reported satisfaction with the app experience | 6-months following trial commencement
  score of patient-reported questionnaire designed to capture the user experience and perceived app functionality using a 5-point Likert scale (from 1 (terrible) to 5 (amazing)). The set of questions pertains to Mobile App User Experience Ratings. Higher scores mean a better outcome.
  Example of question: "On a scale of 1 (terrible) to 5 (amazing), how satisfied are you with the navigation of the app?"
Patient reported satisfaction with communication with the treating physician | 6-months following trial commencement
  score of patient-reported questionnaire designed to capture the confidence in recall or comfort with the physician-patient relationship using a 5-point Likert scale (from 1 (not at all) to 5 (very)). The sets of questions cover the categories: Communicating and Recall at a Consultation, Comfort and Confidence at a Consultation, Relationship with doctor, and Learning. Higher scores mean a better outcome.
  Example of question: "On a scale of 1 (not at all) to 5 (very), how comfortable are you explaining your concern(s), symptoms and goals to your doctor?"

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Zakhari, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- McGill University Health Center, Montreal, Quebec, Canada